CLINICAL TRIAL: NCT01440101
Title: Multicenter Study of BG00002 in Japanese Subjects With RRMS, Consisting of a Multiple-Dose, Open-Label Evaluation of Its Safety, Tolerability, Pharmacokinetics and Pharmacodynamics (Part A) and a Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Evaluation of Safety and Efficacy (Part B)
Brief Title: Natalizumab (BG00002, Tysabri) Study in Japanese Participants With Relapsing-Remitting Multiple Sclerosis (RRMS)
Acronym: Tysabri Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101MS203
Record Dates: First submitted 2011-04-14; First posted 2011-09-26 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Double-blind Natalizumab 300 mg (Experimental): 300 mg IV infusions of natalizumab over 60 minutes every 4 weeks for 20 weeks
  Interventions: Drug: Natalizumab (BG00002)
- Double-blind Placebo (Placebo Comparator): IV infusions of placebo over 60 minutes every 4 weeks for 20 weeks
  Interventions: Drug: Placebo
- Open-label Natalizumab (Experimental): 300 mg IV infusions of natalizumab over 60 minutes every 4 weeks for 20 weeks
  Interventions: Drug: Natalizumab (BG00002)

INTERVENTIONS:
Drug: Natalizumab (BG00002)
  Other Names: Tysabri
  Arms: Double-blind Natalizumab 300 mg; Open-label Natalizumab
Drug: Placebo
  Arms: Double-blind Placebo

SUMMARY:
The primary objective of Part A is to determine the safety and tolerability of natalizumab administered over 24 weeks in Japanese participants with relapsing-remitting multiple sclerosis (MS). The endpoints for this will include assessment of adverse evetns (AEs), changes in laboratory evaluations, vital signs, Expanded Disability Status Scale (EDSS) scores, and changes in physical and neurological examination findings. The secondary objectives of Part A are to characterize the pharmacokinetics (PK) profile and pharmacodynamics (PD) of natalizumab.

The primary objective of Part B is to determine if natalizumab, when compared to placebo, is effective in treating Japanese participants with relapsing-remitting MS, as measured by new active lesions on cranial magnetic resonance imaging (MRI) scans over 24 weeks. New active lesions are the sum of the gadolinium-enhancing (Gd+) lesions and any new or newly-enlarging T2-hyperintense lesions that do not enhance. The primary endpoint is the rate of development of new active lesions over 24 weeks.

Secondary objectives of Part B are to determine over 24 weeks whether natalizumab, when compared to placebo, is effective in reducing the frequency of clinical exacerbations, reducing the number of Gd+ lesions, reducing the number of new or newly-enlarging T2-hyperintense lesions on brain MRI scans, increasing the proportion of relapse-free participants, and improving outcomes on visual analog scale (VAS) assessing the participant's global impression of his/her well-being. Additional objectives are to assess the safety and tolerability, the incidence of serum antibodies to natalizumab and the PK profile of natalizumab.

DETAILED DESCRIPTION:
This multicenter study has 2 parts and is designed to provide data in Japanese participants, as required for registration of natalizumab (BG00002) in Japan. Part A will consist of an open-label cohort of 12 participants who will receive 300 mg natalizumab intravenously (IV) every 4 weeks over a 6-month treatment period. Part B will consist of a double-blind, placebo-controlled cohort of approximately 90 participants randomized in a ratio of 1:1 to receive IV infusions of placebo or 300 mg BG00002 every 4 weeks over a 6-month period.

ELIGIBILITY:
Part A

Key Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law.
* Must have a diagnosis of relapsing-remitting MS, as defined by the revised McDonald criteria 1 through 4 (Polman et al, 2005). All other possible neurologic diagnoses must have been reasonably excluded by means of laboratory and/or imaging studies, in the opinion of the Investigator.
* Japanese men and women aged 18 to 65, inclusive, at the time of informed consent.
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study and be able to continue contraception for 12 weeks after their last dose of study treatment.
* Must have an Expanded Disability Status Scale (EDSS) score between 0.0 and 6.0, inclusive.
* Must have experienced at least 1 medically documented clinical exacerbation within 12 months of enrollment.
* Must be willing to remain free from concomitant immunosuppressive or immunomodulatory treatment (including interferon beta [IFNβ] and chronic systemic corticosteroids) for the duration of the study.
* Must have a baseline MRI, conducted within 35 calendar days prior to enrollment.

Key Exclusion Criteria:

* Diagnosis or history of neuromyelitis optica (NMO), e.g., a long spinal lesion extending over 3 or more vertebral bodies was detected, or the subject has a history of positive tests for anti-aquaporin-4 (anti-AQP4) antibodies.
* The subject is considered by the Investigator to be immunocompromised, based on medical history, physical examination, laboratory testing, or prior immunosuppressive or immunomodulating treatment.
* An MS exacerbation (relapse) within 30 days prior to enrollment or, in the opinion of the Investigator, the subject has not stabilized from a relapse prior to enrollment at Week 0.
* History of malignancy.
* Known history of, or positive test result for human immunodeficiency virus (HIV) infection.
* Known history of or positive test result for hepatitis C virus or hepatitis B virus within the year prior to enrollment.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* A clinically significant infectious illness within 30 days prior to enrollment.
* Abnormal liver function test results at screening: alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >2 times of the upper limit of normal (ULN) or bilirubin >1.5 times of the ULN during screening.
* Previous treatment with natalizumab, any murine protein, or any other therapeutic monoclonal antibody.
* Any prior treatment with any of the following medications: total lymphoid irradiation, cladribine, T-cell or T-cell receptor vaccination.
* Treatment with immunosuppressant medications, e.g., azathioprine, cyclophosphamide, methotrexate, and fingolimod within 6 months prior to enrollment, or mitoxantrone and cyclosporine within 12 months prior to enrollment.
* Treatment with any of the following medications or procedures within 6 months prior to enrollment: intravenous immunoglobulin (IVIg), plasmapheresis, or cytapheresis.
* Treatment with immunomodulatory medications (including IFNβ and glatiramer acetate [GA]) within 2 weeks of enrollment.
* Treatment with any of the following medications within 30 days of enrollment: intravenous corticosteroid treatment, systemic corticosteroid treatment, 4-aminopyridine or related products.
* Participation in any other investigational treatment within the 6 months prior to enrollment or concurrent with this study.

Part B

Key Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law.
* Must have a diagnosis of relapsing-remitting MS, as defined by the revised McDonald criteria 1 through 4 (Polman et al, 2005). All other possible neurologic diagnoses must have been reasonably excluded by means of laboratory and/or imaging studies, in the opinion of the Investigator.
* Japanese men and women aged 18 to 65, inclusive, at the time of informed consent.
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study and be able to continue contraception for 12 weeks after their last dose of study treatment.
* Must have an EDSS score between 0.0 and 5.5, inclusive.
* Must have experienced at least 1 medically documented clinical exacerbation within 12 months of enrollment.
* Must be willing to remain free from concomitant immunosuppressive or immunomodulatory treatment (including IFNβ and chronic systemic corticosteroids) for the duration of the study.
* Prior to enrollment all subjects must have: a screening MRI, or documentation of an MRI within the subject's medical record within 1 year of the screening visit, which reveals 3 or more T2 hyperintense lesions consistent with MS, and a baseline MRI, conducted within 7 calendar days prior to enrollment, which reveals at least 1 MRI lesion consistent with MS.

Key Exclusion Criteria

* Diagnosis or history of NMO, e.g., a long spinal lesion extending over 3 or more vertebral bodies was detected, or the subject has a history of positive tests for anti-AQP4 antibodies.
* The subject is considered by the Investigator to be immunocompromised, based on medical history, physical examination, laboratory testing, or prior immunosuppressive or immunomodulating treatment.
* An MS exacerbation (relapse) within 30 days prior to enrollment or, in the opinion of the Investigator, the subject has not stabilized from a relapse prior to enrollment at Week 0.
* History of malignancy.
* Known history, or positive test result of HIV infection.
* Known history of or positive test result for hepatitis C virus or hepatitis B virus within the year prior to Enrollment.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* A clinically significant infectious illness within 30 days prior to Enrollment.
* Abnormal liver function test results at screening: ALT or AST >2 times of the ULN or bilirubin >1.5 times of the ULN during screening.
* Previous treatment with natalizumab, any murine protein, or any other therapeutic monoclonal antibody.
* Any prior treatment with any of the following medications: total lymphoid irradiation, cladribine, T-cell or T-cell receptor vaccination.
* Treatment with immunosuppressant medications, e.g., azathioprine, cyclophosphamide, methotrexate, and fingolimod within 6 months prior to enrollment, or mitoxantrone and cyclosporine within 12 months prior to enrollment.
* Treatment with any of the following medications or procedures within 6 months prior to enrollment: IVIg, plasmapheresis, or cytapheresis.
* Treatment with immunomodulatory medications (including IFNβ and GA) within 2 weeks of enrollment.
* Treatment with any of the following medications within 30 days of enrollment: intravenous corticosteroid treatment, systemic corticosteroid treatment, 4-aminopyridine or related products.
* Participation in any other investigational treatment within the 6 months prior to enrollment or concurrent with this study.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (17):
- Japan (17):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kawagoe
  - Research Site, Kyoto
  - Research Site, Morioka
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Otaku
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Suita
  - Research Site, Tokorozawa
  - Research Site, Tokyo
  - Research Site, Tsukuba
  - Research Site, Ube
  - Research Site, Yokohama

REFERENCES:
- [Derived] Saida T, Kira JI, Kishida S, Yamamura T, Sudo Y, Ogiwara K, Tibung JT, Lucas N, Subramanyam M; Natalizumab Trial Principal Investigators. Efficacy, safety, and pharmacokinetics of natalizumab in Japanese multiple sclerosis patients: A double-blind, randomized controlled trial and open-label pharmacokinetic study. Mult Scler Relat Disord. 2017 Jan;11:25-31. doi: 10.1016/j.msard.2016.11.002. Epub 2016 Nov 11. PMID 28104251
- [Derived] Saida T, Kira JI, Kishida S, Yamamura T, Ohtsuka N, Dong Q, Tibung JT. Natalizumab for Achieving Relapse-Free, T1 Gadolinium-Enhancing-Lesion-Free, and T2 Lesion-Free Status in Japanese Multiple Sclerosis Patients: A Phase 2 Trial Subanalysis. Neurol Ther. 2017 Jun;6(1):153-159. doi: 10.1007/s40120-016-0062-4. Epub 2017 Jan 11. PMID 28078634

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part, multicenter study, each part (open-label, double-blind) comprising discrete cohorts of BG00002-naïve participants.
Groups:
- Open Label Natalizumab: 300 mg intravenous (IV) infusions of natalizumab (BG00002) over 60 minutes every 4 weeks for 20 weeks
- Double-Blind Natalizumab: 300 mg IV infusions of natalizumab (BG00002) over 60 minutes every 4 weeks for 20 weeks
Period: Overall Study
Arm/Group | Open Label Natalizumab | Double-Blind Placebo | Double-Blind Natalizumab
Started | 12 | 47 | 47
Completed | 10 | 43 | 46
Not Completed | 2 | 4 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This was a 2-part, multicenter study, each part (open-label, double-blind) comprising discrete cohorts of BG00002-naïve participants.
Groups:
- Open Label Natalizumab; Double-Blind Natalizumab: 300 mg IV infusions of natalizumab (BG00002) over 60 minutes every 4 weeks for 20 weeks
- Total: Total of all reporting groups
Arm/Group | Open Label Natalizumab | Double-Blind Placebo | Double-Blind Natalizumab | Total
Number analyzed (Participants) | 12 | 47 | 47 | 106
Age, Customized [Number; unit: participants]
  18 to < 20 years | 0 | 2 | 0 | 2
  20 to < 30 years | 1 | 8 | 9 | 18
  30 to < 40 years | 6 | 24 | 18 | 48
  40 to < 50 years | 3 | 10 | 16 | 29
  50 to < 60 years | 1 | 3 | 3 | 7
  >/= 60 years | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 32 | 34 | 73
  Male | 5 | 15 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events (AEs)
Description: AE=any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. Serious AE (SAE)=any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, was a life threatening event; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; or any other medically important event that, in the opinion of the Investigator, may have jeopardized the participant or may have required intervention to prevent one of the other outcomes listed in the definition above. Events were categorized as related or not related; severity was categorized as mild, moderate, or severe.
Time Frame: Baseline (Week 0) to Week 24
Population: All participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
participants
  Participants with an adverse event (AE) | 8
  Participants with a moderate or severe event | 4
  Participants with a severe event | 1
  Participants with an AE related to study drug | 3
  Participants with a serious event (SAE) | 2
  Participants with an SAE related to study drug | 1
  Participants discontinuing treatment due to an AE | 1
  Participants withdrawing from study due to an AE | 2

2. Primary Outcome: Part B: Rate of Development of New Active Lesions Over 24 Weeks
Description: New active lesions were the sum of the gadolinium-enhancing (Gd+) lesions and any new or newly enlarging T2 hyperintense lesions that did not enhance as seen on cranial magnetic resonance imaging (MRI) scans. The rate is calculated for each participant as the ordinary least squares slope of the cumulative new active lesions over time.
Time Frame: Baseline (Week 0) to Week 24
Population: Missing new Gd+ or new or newly-enlarging, non-enhancing T2 hyperintense lesions were imputed using linear interpolation between the 2 adjacent non-missing values. For participants who discontinued the study, linear interpolation reduced to last observation carried forward (LOCF) was used for imputing any remaining missing values.
Measure: Mean (Standard Deviation); unit: lesions per week over 24 weeks
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
lesions per week over 24 weeks | 0.352 (0.5648) | 0.058 (0.0748)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value obtained from the Mann-Whitney U test stratified by the presence or absence of Gd+ lesions at baseline

3. Secondary Outcome: Part B: Cumulative Number of New Active Lesions Over 24 Weeks
Time Frame: Baseline (Week 0) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
lesions | 8.5 (13.35) | 1.5 (2.06)

4. Secondary Outcome: Part B: Adjusted Annualized Relapse Rate Over 24 Weeks
Description: The frequency of clinical exacerbations over 24 weeks was assessed using an annualized relapse rate that was calculated for each treatment group as the total number of relapses experienced in the group over the 24 weeks of treatment, divided by the total number of subject-years followed in the study. Obtained from a Poisson regression model, adjusted for the baseline relapse rate.
Time Frame: Week 24
Measure: Number (95% Confidence Interval); unit: relapses per year
Units Other Than Participants: Participants with Relapse
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
Number analyzed (Participants with Relapse) | 27 | 9
relapses per year | 1.727 [1.218 to 2.448] | 0.532 [0.286 to 0.992]

5. Secondary Outcome: Part B: Cumulative Number of Gd+ Lesions Over 24 Weeks
Time Frame: Baseline (Week 0) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
lesions | 7.4 (12.15) | 1.2 (1.68)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Test type: Superiority or Other; p < 0.001, Van Elteren test — P-value obtained from the Van Elteren test stratified by the presence or absence of Gd+ lesions at baseline

6. Secondary Outcome: Part B: Cumulative Number Of New Or Newly Enlarging, Non-Enhancing T2-Hyperintense Lesions Over 24 Weeks
Time Frame: Baseline (Week 0) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
lesions | 1.1 (1.84) | 0.3 (0.91)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Test type: Superiority or Other; p = 0.006, Wilcoxon rank sum test

7. Secondary Outcome: Part B: Number of Participants Who Were Relapse Free Over 24 Weeks
Description: Participants were categorized as relapse free=yes, relapse free=no, or relapse free=unknown. The category of relapse free=unknown includes participants who withdrew from the study and did not experience a relapse prior to withdrawal.
Time Frame: Baseline (Week 0) to Week 24
Population: All participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
participants
  Relapse free = yes | 18 | 37
  Relapse free = no | 27 | 9
  Relapse free = unknown | 2 | 1
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Relapse-free proportions compared using a two-sided Fisher exact test. In the analysis, participants with unknown status are considered to have relapsed; Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in proportions = 0.404, 95% CI 2-sided [0.223 to 0.586]

8. Secondary Outcome: Part B: Change From Baseline to Weeks 12 and 24 in the Global Assessment of Well-Being As Assessed by Participants Using a Visual Analog Scale (VAS)
Description: The participant's self-rating of global impression of his/her well-being was assessed with a VAS. The instrument ranged from 0 to 100 (mm), where a score of 0 denoted 'poor' and a score of 100 denoted 'excellent.'
Time Frame: Baseline (Week 0), Week 12, Week 24
Population: n = all participants with an assessment at baseline and given timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
units on a scale
  Baseline; n=47, 47 | 63.5 (23.66) | 69.6 (20.70)
  Change from Baseline at Week 12; n=47, 47 | -4.9 (24.89) | -5.3 (21.49)
  Change from Baseline at Week 24; n=44, 46 | -2.9 (25.20) | -4.8 (17.40)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Change from Baseline to Week 12; Test type: Superiority or Other; p = 0.729, ANCOVA — P-value for comparison between the treated and placebo groups was based on analysis of covariance, adjusted for the baseline VAS score
Statistical Analysis 2: Comparison: Double-Blind Placebo vs Double-Blind Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.942, ANCOVA — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Part A: Concentration of Natalizumab in Serum
Description: The concentration of BG00002 in serum was determined using an Enzyme Linked Immunosorbent Assay (ELISA).
Time Frame: Week 0: pre-dose, post-dose and 2, 24, 48 and 96 hours post-dose; 7, 14, and 21 days post-dose; Weeks 4, 8, 12, and 16: pre-dose; Week 20 pre-dose, post-dose, and 2, 24, 48 and 96 hours post-dose; 7, 14, 21, and 28 days post-dose
Population: Participants who received at least 1 infusion of BG00002 with at least 1 post-baseline assessment of BG00002 serum concentration; n = the number of participants with an assessment at given timepoint. At Weeks 8, 12, and 16, one participant had values less than the lower limit of quantitation (<LLQ) and was not counted in the n for that timepoint.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
µg/mL
  Week 0: pre-dose; n=12 | NA (NA) — All values were below the limit of quantification.
  Week 0: post-dose; n=12 | 119.4550 (18.86145)
  Week 0: 4 hours post-dose; n=12 | 111.8159 (18.35129)
  Week 0: 24 hours post-dose; n=12 | 100.5707 (26.17036)
  Week 0: 48 hours post-dose; n=12 | 92.5144 (18.26611)
  Week 0: 96 hours post-dose; n=12 | 73.2038 (17.02067)
  7 days post-dose; n=12 | 62.3874 (16.49046)
  14 days post-dose; n=12 | 41.2363 (12.02968)
  21 days post-dose; n=12 | 30.9994 (11.45474)
  Week 4: pre-dose; n=12 | 22.5702 (9.55131)
  Week 8: pre-dose; n=11 | 24.7048 (15.50352)
  Week 12: pre-dose; n=10 | 27.9105 (16.06085)
  Week 16: pre-dose; n=10 | 32.9645 (16.41578)
  Week 20: pre-dose; n=10 | 36.2724 (14.51395)
  Week 20: post-dose; n=10 | 145.5353 (38.26877)
  Week 20: 4 hours post-dose; n=10 | 137.6666 (30.47429)
  Week 20: 24 hours post-dose; n=10 | 130.8829 (30.17375)
  Week 20: 48 hours post-dose; n=10 | 120.0772 (28.68860)
  Week 20: 96 hours post-dose; n=10 | 103.3549 (26.94133)
  Week 20: 7 days post-dose; n=10 | 86.2563 (24.70785)
  Week 20: 14 days post-dose; n=10 | 65.7307 (24.60531)
  Week 20: 21 days post-dose; n=10 | 52.4002 (21.41919)
  Week 20: 28 days post-dose; n=10 | 35.8368 (16.33283)

10. Secondary Outcome: Part B: Concentration of Natalizumab in Serum
Description: The concentration of BG00002 in serum was determined using an Enzyme Linked Immunosorbent Assay (ELISA).
Time Frame: Baseline (Week 0), Week 12, Week 24
Population: Randomized participants who received at least 1 infusion of BG00002 and had at least 1 post-baseline assessment of BG00002 serum concentration; n = the number of these participants with an assessment at given timepoint. Participants with values <LLQ were not counted in the n for that timepoint.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Double-Blind Natalizumab
Number analyzed (Participants) | 47
µg/mL
  Baseline; n=47 | NA (NA) — All participants had values < LLQ.
  Week 12; n=45 | 32.6475 (14.68246)
  Week 24; n=45 | 44.4830 (22.53573)

11. Secondary Outcome: Part A: Pharmacokinetic (PK) Profile of Natalizumab in Serum: Cmax
Description: Observed maximum concentration (Cmax) was calculated using non-compartmental methods.
Time Frame: Dose 1/Week 0: pre-dose, post-dose and 4, 24, 48 and 96 hours post-dose; Dose 6/Week 20 pre-dose, post-dose, and 4, 24, 48 and 96 hours post-dose; 7, 14, and 21 days post-dose
Population: Randomized participants who received at least 1 infusion of BG00002 and had at least 1 post-baseline assessment of BG00002 serum concentration; n = the number of these participants with an assessment at given timepoint.
Measure: Geometric Mean (Full Range); unit: µg/mL
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
µg/mL
  Dose 1/Week 0; n=12 | 119.58 [89.4 to 166.0]
  Dose 6/Week 20; n=10 | 144.36 [92.6 to 221.0]

12. Secondary Outcome: Part A: Pharmacokinetic (PK) Profile of Natalizumab in Serum: AUC(0-last) and (0-AUC∞)
Description: Area under the curve to the last measurable concentration (AUC[0-last]); and area under the curve extrapolated to infinity (0-AUC∞) were calculated using non-compartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: µg*h/mL
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
µg*h/mL
  AUC(0-last), Dose 1/Week 0; n=12 | 31574.6 [24462 to 49818]
  AUC(0-last), Dose 6/Week 20; n=10 | 46094.8 [30407 to 71319]
  AUC(0-∞), Dose 1/Week 0; n=12 | 43172.6 [25631 to 68072]

13. Secondary Outcome: Part A: Pharmacokinetic (PK) Profile of Natalizumab in Serum: Tmax and T1/2
Description: Time to maximum concentration (Tmax) and half-life (T1/2) were calculated using non-compartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
hours
  Tmax, Dose 1/Week 0; n=12 | 1.49 [1.0 to 22.0]
  Tmax, Dose 6/Week 20; n=10 | 2.27 [1.0 to 6.0]
  T1/2, Dose 1/Week 0; n=12 | 344.9 [158 to 697]
  T1/2, Dose 6/Week 20; n=10 | 381.2 [181 to 533]

14. Secondary Outcome: Part A: Pharmacokinetic (PK) Profile of Natalizumab in Serum: Vd
Description: Volume of distribution (Vd) was calculated using non-compartmental methods.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
L
  Dose 1/Week 0; n=12 | 3.422 [2.30 to 5.05]
  Dose 6/Week 20; n=10 | 3.561 [2.19 to 6.05]

15. Secondary Outcome: Part A: Pharmacokinetic (PK) Profile of Natalizumab in Serum: CL
Description: Systemic clearance (CL) was calculated using non-compartmental methods.
Time Frame: Dose 1/Week 0: pre-dose, post-dose and 4, 24, 48 and 96 hours post-dose
Population: Randomized participants who received at least 1 infusion of BG00002 and had at least 1 post-baseline assessment of BG00002 serum concentration.
Measure: Geometric Mean (Full Range); unit: mL/h
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
mL/h | 6.9497 [4.410 to 11.700]

16. Secondary Outcome: Part B: Status of Serum Antibodies to Natalizumab
Description: Persistent positivity is defined as 2 positive results separated by at least 6 to 12 weeks.
Time Frame: Baseline (Week 0) and Week 24
Population: Participants with one or more post-baseline screening antibody result.
Measure: Number; unit: participants
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
participants
  Negative at all post-dose results | 47 | 45
  Positive at any time | 0 | 2
  Positive at final evaluation | 0 | 1
  Persistently positive | 0 | 1

17. Secondary Outcome: Part B: Number of Participants With Adverse Events (AEs)
Description: as for outcome 1
Time Frame: Baseline (Week 0) to Week 24
Measure: Number; unit: participants
Arm/Group | Double-Blind Placebo | Double-Blind Natalizumab
Number analyzed (Participants) | 47 | 47
participants
  Participants with an adverse event (AE) | 41 | 34
  Participants with a moderate or severe AE | 30 | 14
  Participants with a severe AE | 5 | 0
  Participants with an AE related to study drug | 7 | 7
  Participants with a serious event (SAE) | 11 | 7
  Participants with an SAE related to study drug | 1 | 1
  Participants discontinuing treatment due to an AE | 1 | 0
  Participants withdrawing from study due to an AE | 1 | 0

18. Secondary Outcome: Part A: Natalizumab Binding Saturation Of α4 Integrin Sites On Peripheral Blood Mononuclear Cells (PBMC)
Description: Pharmacodynamic activity was assessed by measuring the degree of saturation by BG00002 of the very late antigen-4 (VLA-4, also known as α4β1 integrin) receptor on peripheral blood mononuclear cell populations. This was accomplished by staining cells with phycoerythrin-conjugated anti-human immunoglobulin G4 (IgG4) antibody (hIgG4-PE) to label the cell-bound BG00002, followed by flow cytometric detection and quantification.
Time Frame: Pre-dose; 4 hours post-dose; 7, 14, 21, and 28 days post-dose; Weeks 8, 12, and 16: pre-dose; Week 20: pre-dose; 4 hours post-dose; 7, 14, 21, and 28 days post-dose
Population: Participants in Part A who received a dose of BG00002 and had at least 1 post-baseline assessment of α4-integrin saturation; n=participants with an assessment at timepoint.
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
percent saturation
  Pre-dose (n=12) | 6.282 (1.6450)
  4 hours post-dose (n=12) | 88.371 (4.6811)
  7 days post-dose (n=12) | 85.491 (7.1019)
  14 days post-dose (n=12) | 77.929 (6.8396)
  21 days post-dose (n=12) | 71.362 (6.8992)
  28 days post-dose (n=12) | 69.742 (7.3283)
  Week 8: pre-dose (n=11) | 64.057 (20.2412)
  Week 12: pre-dose (n=11) | 60.615 (22.0351)
  Week 16: pre-dose (n=10) | 75.485 (4.4088)
  Week 20: pre-dose (n=10) | 75.314 (7.1022)
  Week 20: 4 hours post-dose (n=10) | 88.859 (5.0230)
  Week 20: 7 days post-dose (n=10) | 83.575 (5.9416)
  Week 20: 14 days post-dose (n=10) | 80.376 (5.4459)
  Week 20: 21 days post-dose (n=10) | 80.842 (5.5828)
  Week 20: 28 days post-dose (n=10) | 70.897 (4.5757)

19. Secondary Outcome: Part A: Summary of Lymphocyte Counts Over Time
Time Frame: Baseline [Week 0]); 28 days post-dose; Weeks 12, 24, and 32 (follow-up)
Population: Participants in Part A who received a dose of BG00002 and had at least 1 post-baseline assessment of lymphocytes; n=participants with assessment at timepoint.
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | Open Label Natalizumab
Number analyzed (Participants) | 12
cells/microliter
  Screening; n=12 | 1708.3 (556.71)
  Pre-dose; n=12 | 1775.0 (534.49)
  28 days Post-dose; n=12 | 3016.7 (845.13)
  Week 12; n=11 | 3018.2 (1112.49)
  Week 24; n=10 | 3340.0 (939.50)
  Week 32 Follow-up; n=2 | 1550.0 (70.71)

ADVERSE EVENTS:
Time Frame: AEs were collected from Baseline (Week 0) through Week 24 (treatment period) + 20 Weeks (or 24 weeks after last infusion). Serious adverse events (SAEs) were collected from the time of informed consent.
Arm/Group | Open Label Natalizumab | Double-Blind Placebo | Double-Blind Natalizumab
Serious Adverse Events (participants affected / at risk) | 2/12 | 11/47 | 7/47
Other Adverse Events (participants affected / at risk) | 8/12 | 32/47 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Natalizumab (N=12) | Double-Blind Placebo (N=47) | Double-Blind Natalizumab (N=47)
Retinal Detachment (Eye disorders) | 1 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 10 | 4
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Asperger's Disorder (Psychiatric disorders) | 0 | 0 | 1
Somatoform Disorder (Psychiatric disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Natalizumab (N=12) | Double-Blind Placebo (N=47) | Double-Blind Natalizumab (N=47)
Nasopharyngitis (Infections and infestations) | 3 | 14 | 9
Cystitis (Infections and infestations) | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 2 | 3
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 3 | 0 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 2 | 17 | 8
Central Nervous System Lesion (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0
Eye Discharge (Eye disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.